CLINICAL TRIAL: NCT00837629
Title: An Open-label Non-interventional Evaluation of Efficacy of Symbicort® Forte Turbuhaler 320/9 µg (Budesonide / Formoterol) and Symbicort® Turbuhaler® 160/4,5 µg (Budesonide / Formoterol)in Functional Status Improvement of Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Evaluation of Symbicort® Turbuhaler® (Budesonide/Formoterol) in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Meta Jeras, Mr Ph, Regulatory and Medical Affairs Manager, AstraZeneca
Other Study IDs: NIS-RSI-SYM-2006/1
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive pulmonary disease; COPD; Symbicort Turbuhaler
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This non-interventional study is to analyse the therapeutic effectiveness in patients with severe COPD following a generally accepted 12-week treatment period with Symbicort Turbuhaler, which could anyhow be shortened or extended at physician's discretion.

ELIGIBILITY:
Inclusion Criteria:

* non pregnant female
* COPD with persistent symptoms in spite of regular bronchodilator therapy
* Naive or fixed combination treated patients including patients already on Symbicort Turbuhaler

Exclusion Criteria:

* Hypersensitivity to budesonide, formoterol or inhaled lactose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients (outpatient or hospitalised) in whom Symbicort Turbuhaler is indicated according to the current Summary of product characteristics (SPC)
Sampling Method: Non-Probability Sample
Enrollment: 743 (Actual)
Dates: Start 2007-02; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Reduction in overall Clinical COPD Questionnaire (CCQ) score | 12 weeks

SECONDARY OUTCOMES:
Patient satisfaction | 12 weeks
Physicians' global clinical impression of the treatment | 12 weeks
Evaluation of smoking habits | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Matjaz Flezar, MD, Principal Investigator — Golnik Hospital